CLINICAL TRIAL: NCT03188029
Title: Effect of Repeated Doses of Etomidate on the Adrenocortical Function
Brief Title: Cortisol Level After Repeated Doses of Etomidate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Kaabachi olfa, professor, University Tunis El Manar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 102/2017
Record Dates: First submitted 2017-06-04; First posted 2017-06-15 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Adrenocortical Abnormality
Keywords: ethomidate adrenocortical insufficiency

STUDY DESIGN:
Intervention Model Description: The aim of this study is to investigate the effect of repeated doses of etomidate on the adrenocortical synthesis of corticosteroids in patients scheduled to electroconvulsive therapy every 2 days for 3 to 4 weeks.
  Anesthesia protocol is standardized with 0.5 mg/kg propofol, 0.3 mg/kg etomidate and 0.5 mg/kg succinylcholine.
  Blood samples for cortisol dosage are performed immediately before the first session, 24 hours after the first session, 24 hours after the third session and 24 hours after the sixth session. All blood samples are performed at 9 AM.
  Samples were analyzed at the end of the recruitment, using the Electrochimiluminescence ECLIA -Cobas - Roche. The normal value are between 6.2-19.4 µg/dL.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adrenocortical function (Experimental): repeated general anesthesia with 0.3 mg/kg etomidate, 0.5 mg/kg propofol and 0.5 mg/kg succinylcholine, every 2 days for 3 to 4 weeks for electroconvulsive therapy.
  Interventions: Diagnostic Test: adrenocortical function

INTERVENTIONS:
Diagnostic Test: adrenocortical function — Blood samples for cortisol dosage are performed and 24 hours after the sixth session. All blood samples are performed at 9 and collected in normal tube.
  Blood samples for glycaemia, sodium, potassium and bicarbonates are performed at the same rate.

SUMMARY:
The aim of this study is to investigate the effect of repeated doses of etomidate on the adrenocortical synthesis of corticosteroids in patients aged 18 to 65, ASA status I to III scheduled to electroconvulsive therapy every 2 days for 3 to 4 weeks.

Anesthesia protocol is standardized with 0.5 mg/kg propofol, 0.3 mg/kg etomidate and 0.5 mg/kg succinylcholine.

Blood samples for cortisol dosage are performed immediately before the first session (baseline cortisol), 24 hours after the first session, 24 hours after the third session and 24 hours after the sixth session. All blood samples are performed at 9 and collected in normal tube.

sample were analysed using the Electrochimiluminescence ECLIA -Cobas - Roche. The normal value are between 6.2-19.4 µg/dL . Sample analysis was performed by a biochemist blinded to clinical detail.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of repeated doses of etomidate on the adrenocortical synthesis of corticosteroids in patients scheduled to electroconvulsive therapy under general anesthesia

Patients aged 18 to 65, ASA status I to III and scheduled to electroconvulsive therapy under general anesthesia every 2 days for 3 to 4 weeks, are included in this prospective observational study. Patients with previously documented adrenocortical insufficiency or under corticosteroid medication are not included Anesthesia protocol is standardized with 0.5 mg/kg propofol, 0.3 mg/kg etomidate and 0.5 mg/kg succinylcholine. Induction of anesthesia is performed after 3 minutes of preoxygenation with 6 l/min fresh gas flow with 100% inspired fraction of oxygen. The patients are maintained in facial mask ventilation until recovery. During the procedure heart rate, non-invasive blood pressure, pulsed oximetry and end tidal carbon dioxyde are monitored.

Blood samples for cortisol dosage are performed immediately before the first session (baseline cortisol = C0), 24 hours after the first session (cortisol after a single dose of etomidate = C1), 24 hours after the third session (cortisol after 3 doses of etomidate = C3) and 24 hours after the sixth session (cortisol after six doses of etomidate = C6). All blood samples are performed at 9 and collected in normal tube.

Blood samples were centrifuged (4000 tours during 10 minutes) and congealed at -20°. All congealed samples were analyzed at the end of the recruitment, using the Electrochimiluminescence ECLIA -Cobas - Roche. The normal value are between6.2-19.4 µg/dL . Sample analysis was performed by a biochemist blinded to clinical detail.

For every end point time, heart rate and blood pressure are noted. Blood samples for glycaemia, sodium, potassium and bicarbonates are performed at the same rate.

End point criteria and statistical analysis:

Delta-1-cortisol is defined as the difference between C0 and C1 Delta-3-cortisol is defined as the difference between C0 and C3 Delta-6-cortisol is defined as the difference between C0 and C6 We planned to enroll 30 patients during the twelve months.

Wilcoxon test for depended data will be used to compare:

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65,
* ASA status I to III
* and scheduled to electroconvulsive therapy under general anesthesia every 2 days for 3 to 4 weeks

Exclusion Criteria:

* previously documented adrenocortical insufficiency
* or under corticosteroid medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
evolution of blood cortisol level | up to one week
  blood cortisal (µg.L) using the Electrochimiluminescence ECLIA -Cobas - Roche. The normal value are between 6.2-19.4 µg/dL

SECONDARY OUTCOMES:
blood glucose | up to one week
  glycaemia (g.L)
blood sodium | up to one week
  sodium (mmol.L)
blood potassium | up to one week
  potassium (mmol.L)
blood bicarbonates | up to one week
  bicarbonates (mmol.L)

CONTACTS AND LOCATIONS:
Overall Officials: RADDAOUI KHAIRREDINE, MD, Study Director — KASSAB ORTHOPEDIC INSTITUTE
Locations (1):
- Razi Hospital, Tunis, La Manouba, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided